CLINICAL TRIAL: NCT01772199
Title: Proof of Mechanism Study to Assess the Potential of GSK239512 to Remyelinate Lesions in Subjects With Relapsing Remitting Multiple Sclerosis
Brief Title: Study to Assess Whether GSK239512 Can Remyelinate Lesions in Subjects With Relapsing Remitting Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 116477
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: GSK239512; remyelination; magnetic resonance imaging; Relapsing Remitting Multiple Sclerosis; Histamine 3 Receptor Antagonist; magnetization transfer ratio
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — GSK239512

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK239512 Arm (Experimental): GSK239512 once daily orally, started at 10 mcg and titrated to the maximum tolerated dose, Up to the highest dose of 80 mcg (10 mcg first week, 20 mcg second week, 40 mcg third week, 80 mcg fourth week) followed by 44 week maintenance treatment period
  Interventions: Drug: GSK239512
- Placebo Arm (Placebo Comparator): Placebo once daily orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK239512 — White to almost white, round tablets. Once daily orally, started at 10 mcg and titrated to the maximum tolerated dose, Up to the highest dose of 80 mcg (10 mcg first week, 20 mcg second week, 40 mcg third week, 80 mcg fourth week) followed by 44 week maintenance treatment period
  Arms: GSK239512 Arm
Drug: Placebo — White to almost white, round tablets. Once daily orally.
  Arms: Placebo Arm

SUMMARY:
This is a randomized, parallel group, placebo-controlled study designed to assess whether GSK239512 can enhance lesion remyelination in subjects with Relapsing Remitting Multiple Sclerosis (RRMS). Subjects with RRMS on stable background treatment with either Avonex (Interferon-beta1a) or Copaxone (Glatiramer Acetate) are eligible to participate. Subjects will be randomized in a 1:1 ratio between placebo and GSK239512, and will continue to be managed with their current standard of care therapy (Copaxone or Avonex). The total treatment period is 48 weeks, including a standard 4 week titration period and 44 week maintenance treatment period (which could be adapted to a 5-week titration and 43 week maintenance period, if needed). Titration doses start at 10 micrograms (mcg) and increase up to 80 mcg (10 mcg first week, 20 mcg second week, 40 mcg third week, 80 mcg fourth week). Subjects will be titrated to the maximum tolerated dose with the objective of titrating to the highest dose (80 mcg GSK239512), whenever possible, based on investigator judgement of tolerability. The post-treatment follow-up period will be a minimum of 2 weeks in duration following the end of treatment at Week 48 or early withdrawal, as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 50 years of age
* Diagnosed with a relapsing-remitting course of multiple sclerosis as defined by the appropriate McDonald criteria at the time of diagnosis.
* Diagnosis of RRMS made within approximately 10 years prior to the screening visit (as documented by year of diagnosis or duration of disease), and No physical manifestations of other forms of Multiple Sclerosis (MS) including signs of progression to secondary progressive MS (SPMS)
* Currently compliant with a stable dose regimen of Avonex (Interferon Beta1a) or Copaxone (Glatiramer Acetate) for management of MS for >= 1 year prior to the screening visit
* The occurrence of at least one of the following (within the year preceding the screen visit AND after >=2 months of stable treatment with Avonex OR Copaxone): a) 1 reported and/or documented relapse, OR b) 1 Gadolinium Enhanced (GdE) lesion on MRI
* Currently neurologically stable, in the investigator's judgment, and not actively experiencing or recovering from a recent relapse at the screening visit
* A Kurtzke Expanded Disability Status Scale (EDSS) score of 1 to 4.5 (inclusive) at the screening visit.
* Must agree not to participate in a clinical study involving another investigational drug or device throughout their participation in this study. Non-interventional study participation is allowed if the time involvement and scheduling will not interfere with compliance in this study in the opinion of the investigator
* A female subject is eligible to enter the study if she is a) Not pregnant or nursing, b) Of non-childbearing potential (i.e. women who have had a hysterectomy, are postmenopausal, which is defined as >2 years without menses [female subjects who have been post-menopausal for <2 years must be confirmed with Follicle Stimulating Hormone and estradiol levels], have both ovaries surgically removed or have current documented tubal ligation); or, c) Of childbearing potential and agrees to use the acceptable methods of birth control, for one month prior to the start of investigational product to 1 month after the last dose of investigational product.
* Informed Consent: Must be competent to understand the information given in the Institutional Review Board (IRB) or Independent Ethics Committee (IEC) approved Informed Consent Form (ICF) and must sign the form prior to the initiation of any study procedures

Exclusion Criteria:

* MRI: Unable to undergo MRI scans (e.g. due to pacemaker, severe claustrophobia, hypersensitivity to contrast media), Lacks adequate venous access for administration of Gd-enhancing agent, or Findings on brain MRI scan indicating any clinically significant brain abnormality other than MS (e.g. damage associated with prior traumatic brain injury)
* Past and Concurrent Medical Conditions: a) History of severe and clinically significant CNS trauma with current sequelae (e.g. traumatic brain injury, spinal cord compression), b) Significant concurrent, uncontrolled medical condition or disease which in the opinion of the investigator could (e.g. significant psychiatric disorder, etc), affect the subjects' safety, impair the subject's reliable participation in the trial, impair the evaluation of the endpoints, or necessitate the use of medication not allowed by this protocol, c) History or presence of myelopathy due to spinal cord compression by disk or vertebral disease or chronic progressive myelopathy, d) Diagnosis of any type epilepsy, e) At risk of suicide, as indicated by: A documented history of attempted suicide or significant suicidal ideation during the 6 months preceding the screening visit, OR If in the investigator's judgment the subject is at risk of a suicide attempt based on the screen visit assessment, including the eC-SSRS, f) Presence of significant and routine sleep disturbance (severe insomnia, nocturnal wandering, confusion, disorientation, agitation, or vivid dreams) that has a negative impact on quality of life that, in the judgement of the investigator, may increase the risk of tolerability issues during dose escalation, g) Presence or history of hallucinations that, in the judgement of the investigator, may increase the safety risk to the subject, h) Known diagnosis or history consistent with positive human immunodeficiency virus (HIV)
* Past and Current Medications and Therapies: Have had treatment with the following to manage their MS: a) Within 1 year: fingolimod (e.g. Gilenya), Rebif (interferon beta1a), interferon beta1b (e.g. Betaseron), mycophenolate mofetil (e.g. CellCept), or Recently approved medication or formulation indicated for the management of MS. Consult with GlaxoSmithKline (GSK) Medical Monitor if there are specific questions regarding eligible treatments b) Within 2 years: natalizumab (e.g. Tysabri), alemtuzumab (e.g. Campath), daclizumab (e.g. Zenapax), rituximab (e.g. Rituxan), mitoxantrone (e.g. Novantrone), cladribine (e.g. Leustatin), or azathioprine (e.g. Imuran)
* Have used corticotropin to manage a relapse within 6 months prior to Screen Visit.
* Have had treatment with the following and were unable to discontinue and refrain from treatment for the specified time period and are not able to discontinue use throughout participation in the clinical trial: dalfampridine /fampridine (e.g. Ampyra) - 1 month prior to Screen Visit, nabiximols (e.g. Sativex) - 1 month prior to Screen Visit, amantadine (e.g. Symmetrel) - 3 months prior to Screen Visit, or leflunomide (e.g. Arava) - 1 year prior to Screen Visit
* Have used the following medications within the last 30 days or 5 half-lives (whichever is longer) prior to screening and are not able to discontinue use throughout participation in the clinical trial: Any CNS stimulants (e.g., modafinil, dexamphetamine, methylphenidate), Known potent P-glycoprotein inhibitors (e.g. itraconazole, ketoconazole, cyclosporin, loperamide, diltiazem, verapamil, spironolactone, quinidine, bepridil, quinine, carvedilol), Known potent inhibitors or inducers of the CYP3A4 enzyme (e.g., verapamil, ketoconazole, cimetidine, rifampin, modafinil), CNS-penetrant antihistamines (e.g. bromopheniramine, chlorpheniramine, clemastine, diphenhydramine, hyrdoxyzine),
* History of medically significant adverse effects (including allergic reactions and hypersensitivities) following treatment with: Histamine H3 receptor antagonist or inverse agonist, Gadolinium enhancing agent, Relapse medication: glucocorticoids (e.g., methylprednisolone) OR A known hypersensitivity to components of the investigational product, relapse medication, or Gadolinium enhancing agent.
* Electrocardiogram (ECG) showing a clinically significant abnormality at screening. Including a QT interval corrected using Bazett's and Fridericia's formulas (QTcB or QTcF) interval of >=450 msec or >=480 msec for patients with a Bundle Branch Block.
* Infectious Disease Status at Screening a) Subjects with no documented record of vaccination against Hepatitis B (primary and secondary immunization and booster) AND a positive test for hepatitis B surface antigen (HBsAg and Hepatitis B Core Antibody [IgM anti-HBc]), b) Subjects with serologic evidence of active Hepatitis C, as indicated by a positive Hepatitis C Virus(HCV) RNA test and anti-HCV antibody test
* Laboratory Values at Screening: Hematology: Total white cell count <2.0 x 109/L, Neutrophils <1.0 x 109/L, Platelets <75 x 109/L (If out of range, platelet count can be repeated to exclude platelet clumping), or Haemoglobin < 80 g/L.
* Screening clinical chemistry liver function test: Alanine aminotransferase (ALT) >2.0 x upper limit of normal (ULN), Aspartate aminotransferase (AST) >2.0 x ULN, Alkaline phosphatise (ALP) >1.5 x ULN, or Bilirubin >1.5 x ULN.
* Documented renal insufficiency or laboratory results indicative of renal insufficiency (due to risks associated with administration of Gadolinium based contrast agents to subjects with moderate to severe kidney disease): Estimated Creatinine Clearance (Cockroft-Gault) <60 mL/minute
* If known, or according to investigator judgement, subject is suspected of not being able to comply with the study protocol requirements. Contributing factors to this assessment by the investigator could be, but not limited to: job demands, substance abuse, alcoholism, drug dependency or psychological disorder
* Prior participation in a clinical trial or use of an investigational product for a non approved intervention: Prior use of an investigational drug for MS or a condition other than MS within 4 weeks or 5 half-lives (whichever is longer) prior to screening. The GSK Medical Monitor should be consulted to confirm eligibility

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 131 (Actual)
Dates: Start 2013-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Mean change in gadolinium (Gd) enhanced (GdE) lesion magnetization transfer ratio (MTR) differences (calibrated to reference scan) from before enhancement to stable recovery (>=3 months post new GdE lesion) | Up to Week 48
  A single Baseline magnetic resonance image (MRI) prior to randomization. Following randomization, a total of 8 MRIs at approximate 6 week intervals: Week 6, Week 12, Week 18, Week 24, Week 30, Week 36, Week 42, Week 48. Reference MRI: In order to accommodate variations in MTR images acquired using different scanners, the images must be normalized to eliminate intensity shifts and contrast variations. For each scanner, images from a normal subject will be obtained and processed to serve as a calibration for each scanner prior to initiating scanning for subjects participating in the study
Mean change in Delta MTR lesion MTR differences (calibrated to reference scan) from before lesion appearance to stable recovery (>=3 months post lesion appearance) | Up to Week 48
  A single Baseline MRI prior to randomization Following randomization, a total of 8 MRIs at approximate 6 week intervals: Week 6, Week 12, Week 18, Week 24, Week 30, Week 36, Week 42, Week 48. Reference MRI: In order to accommodate variations in MTR images acquired using different scanners, the images must be normalized to eliminate intensity shifts and contrast variations. For each scanner, images from a normal subject will be obtained and processed to serve as a calibration for each scanner prior to initiating scanning for subjects participating in the study

SECONDARY OUTCOMES:
Change from baseline in T2 lesion MTR at Week 48 | Baseline and Week 48
Cumulative new and enlarging Gd enhancing, T2 and Combined Unique Active lesions comparing placebo to GSK239512 treated subjects | Up to Week 48
Change from baseline at Week 48 in total brain volume, white matter volume and grey matter volume comparing placebo to GSK239512 treated subjects | Baseline and Week 48
Cumulative number of persistent black holes and new unenhancing T1 lesion counts comparing placebo to GSK239512 treated subjects over treatment duration up to Week 48 | Up to Week 48
Proportion of new GdE lesions evolving into chronic (unenhancing) T1 lesions (black holes) comparing placebo to GSK239512 treated subjects over treatment duration up to Week 48 | Up to Week 48
Mean change from baseline in overall cognitive impairment and cognitive domains comparing placebo to GSK239512 treated subjects | Baseline and Week 48
  A cognitive battery (computerized battery) is included in this study to assess the impact, if any, on several cognitive functional domains. The battery will be executed twice during the screen visit to familiarize the subject with the use of the tool
Comparison of Relapse Rates between placebo and GSK239512 treated subjects | Up to 50 Weeks
  A relapse in this protocol is defined as: "patient-reported symptoms or objectively observed signs typical of an acute inflammatory demyelinating event in the central nervous system (CNS), current or historical". It must occur in the absence of fever or infection and should - follow improvement from a previous relapse, occur at least 30 days following the onset of a previous relapse, and be persistent for at least 24 hours
Comparison of Time to First Relapse between placebo and GSK239512 | Up to 50 Weeks
  A relapse in this protocol is defined as: "patient-reported symptoms or objectively observed signs typical of an acute inflammatory demyelinating event in the central nervous system (CNS), current or historical". It must occur in the absence of fever or infection and should - follow improvement from a previous relapse, occur at least 30 days following the onset of a previous relapse, and be persistent for at least 24 hours
Comparison of the proportion of subjects Relapse Free between placebo and GSK239512 treated subjects | Up to 50 Weeks
  A relapse in this protocol is defined as: "patient-reported symptoms or objectively observed signs typical of an acute inflammatory demyelinating event in the central nervous system (CNS), current or historical". It must occur in the absence of fever or infection and should - follow improvement from a previous relapse, occur at least 30 days following the onset of a previous relapse, and be persistent for at least 24 hours
Proportion of subjects with sustained worsening of Expanded Disability Severity Scale (EDSS) over 3 months comparing placebo to GSK239512 treated subjects | Up to 48 Weeks
  The EDSS is an assessment of disability specifically associated with Multiple Sclerosis. The assessment will be captured in the medical records including the detailed assessment and scoring for each functional system and domain
Mean change from baseline in the EDSS functional systems and a subset of component assessments comparing placebo to GSK239512 treated subjects | Up to 48 Weeks
  The EDSS is an assessment of disability specifically associated with Multiple Sclerosis. The assessment will be captured in the medical records including the detailed assessment and scoring for each functional system and domain
Safety and tolerability as assessed by frequency and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Week 50
Safety and tolerability as assessed by percentage of subjects withdrawing due to AEs | Up to Week 50
Safety and tolerability as assessed by summary of suicide behavior and ideation risk as assessed by the electronic Columbia Suicide Severity Rating Scale (eC-SSRS) | Up to Week 50
Safety and tolerability as assessed by summary of suicide behavior and ideation risk as assessed by Possible Suicidality Related Adverse Event (PSRAE) | Up to Week 50
Safety and tolerability as assessed by change from baseline in clinical chemistry, hematology, and urinalysis parameters | Up to Week 50
Safety and tolerability as assessed by frequency of clinical chemistry, hematology, and urinalysis parameters of potential clinical concern | Up to Week 50
Safety and tolerability as assessed by change from baseline in blood pressure | Up to Week 50
Safety and tolerability as assessed by change from baseline in heart rate | Up to Week 50
Safety and tolerability as assessed by change from baseline in Electrocardiogram (ECG) parameters | Up to Week 50
Safety and tolerability as assessed by frequency of vital signs and ECG parameters of potential clinical concern | Up to Week 50
Trough concentration of GSK239512 at Week 4, Week 24, Week 36 and Week 48 | Up to 48 weeks
Sparse Pharmacokinetics (PK) sampling for concentration of GSK239512 at Week 8 | Pre-dose, and 30 minutes (15 min to 1 hour), 2 hours (1 to 4 hours) and 6 hours (4 to 8 hours) post dose
  1 pre-dose and 3 post-dose samples. No samples should be collected within 30 minutes of the previous sample

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (35):
- GSK Investigational Site, Sofia, Bulgaria
- Canada (5):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Gatineau, Quebec
  - GSK Investigational Site, Montreal, Quebec
- Czechia (3):
  - GSK Investigational Site, Jihlava
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Teplice
- Germany (9):
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Alzenau in Unterfranken, Bavaria
  - GSK Investigational Site, Unterhaching, Bavaria
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Berlin, State of Berlin
- Spain (5):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Majadahonda (Madrid)
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Seville
- GSK Investigational Site, Stockholm, Sweden
- Ukraine (8):
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Ivano-Frankivsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Lutsk
  - GSK Investigational Site, Lviv
  - GSK Investigational Site, Poltava
  - GSK Investigational Site, Vinnitsa
- United Kingdom (3):
  - GSK Investigational Site, London
  - GSK Investigational Site, Romford
  - GSK Investigational Site, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 116477 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116477 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116477 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116477 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116477 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116477 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116477 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register